CLINICAL TRIAL: NCT03828448
Title: A Phase II Study Evaluating the Safety and Efficacy of Umbralisib (TGR-1202) in Combination With Ublituximab in Patients With Treatment Naïve Follicular Lymphoma and Small Lymphocytic Lymphoma
Brief Title: Study to Assess Umbralisib Plus Ublituximab in Participants With Treatment Naïve Follicular Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic/Business Decision
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTX-TGR-203
Record Dates: First submitted 2019-01-31; First posted 2019-02-04 (Actual); Results first posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Follicular Lymphoma; Small Lymphocytic Lymphoma
Keywords: Treatment naïve
MeSH Terms: conditions — Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ublituximab; umbralisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ublituximab + Umbralisib (Experimental): Participants were administered ublituximab, 900 milligrams (mg), intravenous (IV) infusion through Cycles 1-6, Cycles 9 and 12. Participants also received umbralisib, 800 mg, oral tablet, daily through Cycles 1-24. 1 Cycle = 28 days.
  Interventions: Drug: Ublituximab; Drug: Umbralisib

INTERVENTIONS:
Drug: Ublituximab — - anti-CD 20 monoclonal antibody administered via IV infusion
  Other Names: TG-1101
Drug: Umbralisib — - PI3K Delta Inhibitor oral daily dose
  Other Names: TGR-1202

SUMMARY:
This is a phase 2, open label study to assess umbralisib in combination with ublituximab in participants with treatment naïve Follicular Lymphoma (FL) and Small Lymphocytic Lymphoma (SLL).

DETAILED DESCRIPTION:
The study will assess the safety and efficacy of umbralisib in combination with ublituximab in participants with treatment naïve FL and SLL. Ublituximab will be administered through Cycle 12, while umbralisib will be administered through Cycle 24. After this time, participants will be followed for progression free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of FL or SLL.
* Measurable disease that requires treatment
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1

Exclusion Criteria:

* Currently or previously received treatment for their lymphoma
* Received wide field radiotherapy within 28 days or limited field radiation within 14 days of Cycle 1 Day 1
* Evidence of hepatitis B virus, hepatitis C virus or known human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - TG Therapeutics Investigational Trial Site, Fort Myers, Florida
  - TG Therapeutics Investigational Trial Site, St. Petersburg, Florida
  - TG Therapeutics Investigational Trial Site, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 34 participants were enrolled at 3 investigative sites in the United States from 10 July 2019 to 31 May 2022.
Period: Overall Study
Arm/Group | Ublituximab + Umbralisib
Started | 34
Completed | 0
Not Completed | 34
Not completed — Sponsor's Discretion | 34

BASELINE CHARACTERISTICS:
Groups:
- Ublituximab + Umbralisib: Participants were administered ublituximab, 900 mg, IV infusion through Cycles 1-6, Cycles 9 and 12. Participants also received umbralisib, 800 mg, oral tablet, daily through Cycles 1-24. 1 Cycle = 28 days.
Arm/Group | Ublituximab + Umbralisib
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 70 [42 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as sum of participants with partial responses (PR) and complete responses (CR). CR was defined as complete disappearance of all evidence of disease and disease-related symptoms. PR was defined as regression of measurable disease and no new sites of disease. Regression= ≥ 50% decrease in sum of the products of diameters (SPD) of index lesions, with no unequivocal increase in size of other lymph nodes, liver, or spleen.
Time Frame: Up to 22 months
Population: Data for this outcome measure was not collected or analyzed as planned as the study was terminated due to sponsor's business decision.
Arm/Group | Ublituximab + Umbralisib
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the interval from Cycle 1/Day 1 to the earlier of the first documentation of definitive disease progression or death from any cause. Appearance of any new lesion more than 1.5 cm in any axis, even if other lesions were decreasing in size was considered relapsed or progressive disease. At least a 50% increase from nadir in one of the following: SPD of index lesions, greatest transverse diameter (GTD) of any individual previously involved node, or GTD of any previously involved node provided that the GTD of that node was ≥ 1.5 cm.
Time Frame: Up to approximately 35 months
Population: as for outcome 1
Arm/Group | Ublituximab + Umbralisib
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE) as Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0
Description: An adverse event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. A TEAE is an AE that starts or worsens after receiving study drug.
Time Frame: Up to approximately 35 months
Population: as for outcome 1
Arm/Group | Ublituximab + Umbralisib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: No safety data was collected and analyzed as planned at the end of study
Description: Study was terminated due to sponsor's business decision. Hence, no safety data was collected and analyzed as planned at the end of study.
Groups:
- Ublituximab + Umbralisib: Participants were administered ublituximab, 900 mg, IV infusion on Days 1, 8, and 15 in Cycle 1 and Day 1 of Cycles 2-6, Cycle 9 and 12. Participants also received umbralisib, 800 mg, oral tablet, daily through Cycles 1-24. 1 Cycle = 28 days.
Arm/Group | Ublituximab + Umbralisib
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Due to sponsor's business decision, the clinical trial was terminated by the sponsor prematurely. No analysis was done at the termination of the trial, therefore, outcome, and safety data are not available and the numbers of participants analyzed are reported as "0."

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT03828448/Prot_SAP_000.pdf